CLINICAL TRIAL: NCT05573230
Title: A Phase 1, Open-Label, Drug Interaction Study to Investigate the Effect of Multiple Doses of Cyclosporine on the Pharmacokinetics of LY3502970 in Healthy Participants
Brief Title: A Drug Interaction Study of Cyclosporine and LY3502970 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18506; J2A-MC-GZGL (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; orforglipron; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam + LY3502970 (Experimental): Midazolam administered orally followed by LY3502970 given orally.
  Interventions: Drug: Midazolam; Drug: LY3502970
- Cyclosporine + Midazolam + LY3502970 (Experimental): Cyclosporine administered in combination with midazolam and LY3502970 given orally.
  Interventions: Drug: Midazolam; Drug: LY3502970; Drug: Cyclosporine

INTERVENTIONS:
Drug: Midazolam — Administered orally.
Drug: LY3502970 — Administered orally.
Drug: Cyclosporine — Administered orally.
  Arms: Cyclosporine + Midazolam + LY3502970

SUMMARY:
The main purpose of this study is to determine the levels of study drug called LY3502970 in the blood stream when administered alone and in combination with cyclosporine in healthy participants. The study will also evaluate the safety and tolerability of LY3502970 in healthy participants. This study will last up to approximately 76 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Participants with a body weight of 45 kilograms (kg) or more and body mass index (BMI) within the range of 18.5 to 35.0 kilograms per meter squared (kg/m²)
* Participants who have a hemoglobin level of at least 11.4 grams/deciliter (g/dL) for female participants and at least 12.5 g/dL for male participants
* Male participants who agree to use highly effective/effective methods of contraception and female participants not of childbearing potential

Exclusion Criteria:

* Participants who have a significant history of or current cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Participants who regularly use known drugs of abuse
* Women who are lactating and who are of child-bearing potential
* Participants who have known allergies to LY3502970, related compounds, or any components of the formulation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3502970 | Predose up to 96 hours postdose
  PK: AUC of LY3502970
PK: Maximum Observed Concentration (Cmax) of LY3502970 | Predose up to 96 hours postdose
  PK: Cmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No